CLINICAL TRIAL: NCT06499233
Title: Efficacy and Safety of Prophylactic Treatment for Pneumocystis Jirovecii Pneumonia (PJP) in Patients With Autoimmune Inflammatory Rheumatic Disease (AIIRD)
Brief Title: Efficacy and Safety of Prophylactic Treatment for Pneumocystis Jirovecii Pneumonia in Patients With Autoimmune Inflammatory Rheumatic Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lingli Dong, Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TJ-IRB20231250
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pneumonia, Pneumocystis; Autoimmune Inflammatory Rheumatic Disease; Autoimmune Diseases; Connective Tissue Disease; Prevention
MeSH Terms: conditions — Pneumonia, Pneumocystis; Autoimmune Diseases; Connective Tissue Diseases | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- TMP/SMX (with PJP high risk) (Experimental): AIIRD patients who have PJP high risk and receive prophylactic Trimethoprim/ Sulfamethoxazole (TMP/SMZ) treatment; Drug intervention: Patients receive Trimethoprim/Sulfamethoxazole (TMP/SMX) 480 mg p.o. every day as PJP Prophylaxis.
  Interventions: Drug: Trimethoprim/Sulfamethoxazole
- no TMP/SMX (with PJP high risk) (No Intervention): AIIRD patients who have PJP high risk and do not receive prophylactic Trimethoprim/ Sulfamethoxazole (TMP/SMZ) treatment.
- TMP/SMX (with PJP low-risk) (Experimental): AIIRD patients who have PJP low risk and receive prophylactic Trimethoprim/ Sulfamethoxazole (TMP/SMZ) treatment; Drug intervention: Patients receive Trimethoprim/Sulfamethoxazole (TMP/SMX) 480 mg p.o. every day as PJP Prophylaxis.
  Interventions: Drug: Trimethoprim/Sulfamethoxazole
- no TMP/SMX (with PJP low-risk) (No Intervention): AIIRD patients who have PJP low risk and do not receive prophylactic Trimethoprim/ Sulfamethoxazole (TMP/SMZ) treatment.

INTERVENTIONS:
Drug: Trimethoprim/Sulfamethoxazole — Patients received Trimethoprim/Sulfamethoxazole (TMP/SMX) 480 mg p.o. every day as PJP Prophylaxis; Treatment duration: at least 28 days, adjusted by the clinician based on the severity of the patient's condition, the patient's tolerance to the drug and treatment willingness).
  Other Names: TMP/SMX
  Arms: TMP/SMX (with PJP high risk); TMP/SMX (with PJP low-risk)

SUMMARY:
This is an open-labeled, prospective clinical study aims at collecting and analyzing baseline characteristics of autoimmune inflammatory rheumatic disease (AIIRD) patients receiving sulfanilamide for preventive purposes, as well as subsequent follow-up data, in order to assess the efficacy and safety of the medication. Additionally, through a stratified analysis of risk factors, the investigators aim to identify the AIIRD population that would benefit most from preventive medication based on a favorable benefit-risk ratio.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was diagnosed with AIIRD according to the International Classification of Diseases and had received steroids or immunosuppressive therapy;
2. The patient had not received standard PJP treatment before enrollment, including the first-line treatment drug TMP/SMZ, or other second-line treatment drugs (including Pentamidine, Atorvastatin, Caspofungin, etc.);
3. The patient was at least 18 years old at the time of enrollment;

Exclusion Criteria:

1. Serious health problems or diseases, including (but not limited to) the following: severe liver damage (ALT, AST elevated above normal value by more than 5 times), severe renal insufficiency (GFR < 30mL/min or Scr > 445umol/L), severe myelosuppression (Hb < 65g/L, PLT < 25×10^9/L or neutrophils < 0.5×10^9/L);
2. Screening test indicates infection with human immunodeficiency virus (HIV), history of lymphomatous hyperplasia of the lymphatic tissue or any malignant tumor of any organ system within the past 5 years, or history of organ transplantation;
3. Participants with a history of allergy to sulfonamide drugs, megaloblastic anemia due to folate deficiency;
4. Pregnant and lactating women;
5. Any medical or psychological condition that the investigator believes would interfere with the participant's ability to comply with the protocol or complete the study;
6. Patients who refuse to comply with the requirements of this study and complete the study;
7. Any other situation that the investigator considers unsuitable for participation in the study (for reasons including but not limited to management reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 800 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with PJP infection | 6 months, 12 months
  Defined as documentation/diagnosis of Pneumocystis from a properly obtained specimen (induced sputum, bronchoalveolar lavage, or biopsy) in a patient with clinical manifestations compatible with PJP.

SECONDARY OUTCOMES:
TMP/SMZ related adverse drug reactions | 6 months, 12 months
  Symptoms and signs that may be related to adverse drug reactions during treatment (such as nausea, vomiting, anorexia, jaundice, rashes and hives, and shock); incidence, duration and severity of adverse events
PJP-related mortality | 6 months, 12 months
  PJP-related mortality at the end of month 6.
All cause mortality | 6 months, 12 months
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Lingli Dong, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT06499233/Prot_ICF_000.pdf